CLINICAL TRIAL: NCT00294671
Title: The Effect of Diflunisal on Familial Amyloidosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, John L. Berk, Principal Investigator, Boston University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS051306 (NIH); FD R 002532 (Other Grant/Funding Number: FDA Office of Orphan Products Development (OOPD)); R01NS051306 (NIH)
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-01

CONDITIONS: Familial Amyloid Polyneuropathy; Familial Amyloidosis
Keywords: familial amyloid polyneuropathy; familial amyloidosis; diflunisal; amyloidosis; transthyretin; peripheral neuropathy; autonomic neuropathy; amyloid cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis, Familial; Amyloidosis; Peripheral Nervous System Diseases | interventions — Diflunisal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diflunisal (Active Comparator): Diflunisal 250 mg po bid
  Interventions: Drug: diflunisal
- Placebo (Placebo Comparator): Placebo 1 po bid
  Interventions: Other: placebo

INTERVENTIONS:
Drug: diflunisal — given twice daily for 24 months
  Arms: Diflunisal
Other: placebo — an inactive substance given twice daily for 24 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if diflunisal can prevent progressive lower leg nerve damage in patients with familial amyloidosis polyneuropathy.

Funding Source - FDA Office of Orphan Products Development (OOPD); National Institute of Neurological Disorders and Stroke (NINDS)

DETAILED DESCRIPTION:
Familial amyloidosis polyneuropathy (FAP) is a rare, lethal, autosomal dominant, neurodegenerative disease characterized by misfolding of variant transthyretin tetramer (TTR) - a transport protein produced by the liver. The disease causes TTR to become unstable, triggering amyloid fibrils to form and leading to peripheral and autonomic nerve dysfunction.

Currently, the only treatment for FAP is a liver transplant, which is expensive and risk-filled. Medicines are needed to treat this disease. Previous in vitro (in a test tube) studies have shown that a common anti-inflammatory drug called diflunisal stabilizes TTR, preventing the formation of amyloid fibrils.

The goal of this 2-year randomized, double-blind, placebo-controlled research study is to establish whether diflunisal can stop the nerve damage, or peripheral neuropathy, resulting from amyloid production in patients with FAP. Scientists already know that diflunisal prevents formation of amyloid in the test tube. This study will determine if the drug can block amyloid production in FAP patients.

Participants will be randomly chosen to receive either diflunisal or an inactive (placebo) pill twice daily for 24 months. Participants will be carefully monitored through 7 follow-up visits, either at the study center or with individual primary care physicians. Participating in the study does not preclude patients from being listed for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* Biopsy proven amyloidosis
* Genotyping of variant transthyretin
* Signs of peripheral or autonomic neuropathy

Exclusion Criteria:

* Use of other non-steroidal anti-inflammatory drugs
* Other causes of sensorimotor polyneuropathy
* Anticipated survival <2 years or liver transplantation in <1 yr
* Liver transplantation
* Profound nerve, heart or kidney impairment
* Pregnancy or unwillingness to use contraception by women of childbearing age
* Active or recent gastrointestinal bleeding
* Non-steroidal or aspirin drug allergy/hypersensitivity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L. Berk, MD, Principal Investigator — Boston University
Locations (8):
- United States (3):
  - Amyloidosis Center, Boston Medical Center, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mount Sinai School of Medicine, Department of Medicine, New York, New York
- IRCCS Policlinico San Matteo, Pavia, Italy
- Japan (2):
  - Kumamoto University, Kumamoto
  - Shinshu University, Matsumoto
- Umea University Hospital, Umeå, Sweden
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
A manuscript analyzing cardiac outcomes is being prepared. We will consider IPD after the manuscript is complete and accepted.

REFERENCES:
- [Derived] Berk JL, Suhr OB, Obici L, Sekijima Y, Zeldenrust SR, Yamashita T, Heneghan MA, Gorevic PD, Litchy WJ, Wiesman JF, Nordh E, Corato M, Lozza A, Cortese A, Robinson-Papp J, Colton T, Rybin DV, Bisbee AB, Ando Y, Ikeda S, Seldin DC, Merlini G, Skinner M, Kelly JW, Dyck PJ; Diflunisal Trial Consortium. Repurposing diflunisal for familial amyloid polyneuropathy: a randomized clinical trial. JAMA. 2013 Dec 25;310(24):2658-67. doi: 10.1001/jama.2013.283815. PMID 24368466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between May 2006 and December 2010 from amyloid centers of excellence in Sweden (Umea), Italy (Pavia), United Kingdom (London), Japan (Matsumoto and Kumamoto), and the United States (New York, Minnesota, and Massachusetts).
Pre-assignment Details: All enrolled participants were randomized to treatment groups.
Groups:
- Diflunisal: Diflunisal 250 mg taken by mouth twice daily for 24 months
- Placebo: Placebo, an inactive substance, taken by mouth twice daily for 24 months
Period: Overall Study
Arm/Group | Diflunisal | Placebo
Started | 64 | 66
Completed | 37 | 26
Not Completed | 27 | 40
Not completed — Lack of Efficacy | 11 | 23
Not completed — Liver transplant | 7 | 9
Not completed — Drug related adverse event (AE) | 4 | 2
Not completed — Non-drug related AE | 3 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Non-compliance | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diflunisal | Placebo | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.7) | 59.2 (12.2) | 59.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 43 | 44 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 52 | 50 | 102
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 69
  United Kingdom | 3 | 4 | 7
  Italy | 10 | 11 | 21
  Japan | 5 | 4 | 9
  Sweden | 12 | 12 | 24
NIS+7 score [Mean (Standard Deviation); unit: units on a scale] — Higher scores indicating greater neurologic deficits (0=no neurologic impairment, 270=no detectable peripheral neurologic function)
  units on a scale | 51.6 (42.8) | 59.0 (50) | 55.3 (46.5)
Kumamoto score [Mean (Standard Deviation); unit: units on a scale] — Higher scores indicating greater neurologic and end organ deficits (0=no neurologic deficits, 102=no detectable peripheral neurologic function)
  units on a scale | 15.3 (10.8) | 16.7 (13.5) | 16.0 (12.2)
Modified BMI [Mean (Standard Deviation); unit: kg/M2 x g/L] — The product of BMI and serum albumin (g/L). Lower scores indicate worse nutritional status.
  kg/M2 x g/L | 1024.4 (226.3) | 1019 (255) | 1021.7 (240.4)
SF-36 physical component score [Mean (Standard Deviation); unit: units on a scale] — Higher scores indicate greater physical quality of life, scale from 0 to 100 points
  units on a scale | 35.9 (11.6) | 34.8 (11) | 35.4 (11.3)
SF-36 mental component score [Mean (Standard Deviation); unit: units on a scale] — Higher scores indicate greater mental quality of life, scale 0-100 points
  units on a scale | 46.6 (14.1) | 46.5 (11.8) | 46.6 (12.9)

OUTCOME MEASURES:

1. Primary Outcome: Neurologic Impairment Score + 7 (NIS+7)
Description: The primary endpoint, the difference in polyneuropathy progression between treatments, was measured by the Neuropathy Impairment Score plus 7 nerve tests (NIS+7) which ranges from 0 (no neurologic deficits) to 270 points (no detectable peripheral nerve function).
Time Frame: Baseline, 1 and 2 years
Population: Longitudinal analysis examined data from all 130 participants using intention-to-treat principles.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Diflunisal | Placebo
Number analyzed (Participants) | 64 | 66
units on a scale
  Change from baseline to 2 years | 8.2 [2.9 to 13.6] | 26.3 [20.2 to 32.4]
  Change from baseline to 1 year | 6.2 [2.8 to 9.6] | 12.5 [8.6 to 16.4]
Statistical Analysis 1: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in NIS+7 change from baseline to 2 years; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in NIS+7 change from baseline to 1years; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

2. Secondary Outcome: Kumamoto Neurologic Scale;
Description: Change from baseline of the Kumamoto Score (0-102 points, increasing with disease severity), a clinical neurologic scale of motor, sensory, and autonomic function combined with heart and kidney end organ measures developed to track disease progression in Familial Amyloid Polyneuropathy (ATTR-FAP)
Time Frame: Baseline, 1 and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Diflunisal | Placebo
Number analyzed (Participants) | 64 | 66
units on a scale
  Change from baseline to 2 years | 3.1 [1.1 to 5.1] | 8.0 [5.8 to 10.3]
  Change from baseline to 1 year | 1.9 [0.1 to 3.7] | 4.1 [2.1 to 6.2]
Statistical Analysis 1: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in Kumamoto score change from baseline to 2 years; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 2: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in Kumamoto score change from baseline to 1 year; Test type: Superiority or Other; p = 0.10, t-test, 2 sided

3. Secondary Outcome: Modified Body Mass Index (mBMI);
Description: The product of body mass index (BMI) and serum albumin level (g/L) [kg/M2xg/L].
Time Frame: Baseline, 1 and 2 years
Measure: Mean (95% Confidence Interval); unit: kg/M2xg/L
Arm/Group | Diflunisal | Placebo
Number analyzed (Participants) | 64 | 66
kg/M2xg/L
  Change from baseline to 2 years | -33.7 [-69.3 to 1.8] | -67.9 [-108.1 to -27.7]
  Change from baseline to 1 year | -18.7 [-51.6 to 14.1] | -38.5 [-74.9 to -2.1]
Statistical Analysis 1: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in mBMI change from baseline to 2 years; Test type: Superiority or Other; p = 0.21, t-test, 2 sided
Statistical Analysis 2: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in mBMI change from baseline to 1 year; Test type: Superiority or Other; p = 0.43, t-test, 2 sided

4. Secondary Outcome: Quality of Life Questionnaire: SF-36 Physical Component Score
Description: The 36 item short-form health survey (SF-36) was used to assess the difference between treatment groups for change of physical component scores over 2 years treatment. Range 0-100; lower scores reflect lower quality-of-life.
Time Frame: Baseline, 1 and 2 years
Population: Longitudinal analysis examined data from all 130 participants using intention-to-treat principles.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Diflunisal | Placebo
Number analyzed (Participants) | 64 | 66
units on a scale
  Change from baseline to 2 years | 1.2 [-1.2 to 3.7] | -4.9 [-7.6 to -2.1]
  Change from baseline to 1 year | 0.7 [-1.1 to 2.5] | -1.9 [-3.9 to 0.2]
Statistical Analysis 1: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in SF-36 physical component change from baseline to 2 years; Test type: Superiority or Other; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in SF-36 physical component change from baseline to 1 year; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

5. Secondary Outcome: Quality of Life Questionnaire: SF-36 Mental Component Score
Description: The 36 item short-form health survey (SF-36) was used to assess the difference between treatment groups for change of mental component scores over 2 years treatment. Range 0-100; lower scores reflect lower quality-of-life.
Time Frame: Baseline, 1 and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Diflunisal | Placebo
Number analyzed (Participants) | 64 | 66
units on a scale
  Change from baseline to 2 years | 3.5 [0.4 to 6.7] | -0.9 [-4.4 to 2.5]
  Change from baseline to 1 year | 2.5 [0.0 to 5.1] | 0.8 [-2.0 to 3.6]
Statistical Analysis 1: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in SF-36 mental component change from baseline to 2 years; Test type: Superiority or Other; p = 0.06, t-test, 2 sided
Statistical Analysis 2: Comparison: Diflunisal vs Placebo; Longitudinal analysis of the difference between placebo and diflunisal treatment groups in SF-36 mental component change from baseline to 1 year; Test type: Superiority or Other; p = 0.37, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 years or until study withdrawal.
Description: Adverse events were collected and analyzed by affected organ system.
Arm/Group | Diflunisal | Placebo
Serious Adverse Events (participants affected / at risk) | 3/64 | 4/66
Other Adverse Events (participants affected / at risk) | 29/64 | 27/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diflunisal (N=64) | Placebo (N=66)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (3) | 2 (3)
Infections and infestations (Infections and infestations) | 0 (0) | 1 (1)
Cardiac disorders (Cardiac disorders) | 2 (2) | 1 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diflunisal (N=64) | Placebo (N=66)
Infections (Infections and infestations) | 24 | 27
GI disorders (Gastrointestinal disorders) | 23 | 25
Nervous system disorders (Nervous system disorders) | 23 | 20
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 19 | 8
General disorders (General disorders) | 19 | 7
Cardiac disorders (Cardiac disorders) | 15 | 9
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 13 | 9
Investigations (Investigations) | 11 | 11
Renal and urinary disorders (Renal and urinary disorders) | 10 | 12
Vascular disorders (Vascular disorders) | 11 | 7
Eye disorders (Eye disorders) | 8 | 9
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 | 9
Psychiatric disorders (Psychiatric disorders) | 5 | 7
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 6 | 6
Surgical and medical procedures (Surgical and medical procedures) | 5 | 3
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 | 3
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 1
Endocrine disorders (Endocrine disorders) | 1 | 0
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 0
Immune system disorders (Immune system disorders) | 1 | 0
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No